CLINICAL TRIAL: NCT04252456
Title: seconD-line Folfiri/aflIbercept in proSpecTIvely Stratified, Anti-EGFR resistaNt, Metastatic coloreCTal Cancer patIents With RAS Validated Wild typE Status
Brief Title: Folfiri/aflIbercept in Metastatic coloreCTal Cancer patIents With RAS Validated Wild typE Status
Acronym: DISTINCTIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-002219-33
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — aflibercept; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Biologically enriched phase II clinical trial. All patients will receive aflibercept in combination with FOLFIRI according to the Italian label.
Masking Description: All patients will receive aflibercept in combination with FOLFIRI according to the Italian label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- standard chemotherapy for advanced colorectal cancer (Other): All patients will receive aflibercept in combination with FOLFIRI according to the Italian label.
  Interventions: Procedure: Aflibercept, 5fluorouracil, Folinic Acid andIrinotecan

INTERVENTIONS:
Procedure: Aflibercept, 5fluorouracil, Folinic Acid andIrinotecan — All patients will receive aflibercept in combination with FOLFIRI according to the Italian label

SUMMARY:
The study will a be a biologically enriched, prospectively stratified phase II trial in RAS wild type metastatic colorectal cancer patients progressing after first-line treatment with oxaliplatin, fluoropyrimidines and an anti-EGFR monoclonal antibody.

All patients will receive aflibercept in combination with FOLFIRI according to the Italian label.

DETAILED DESCRIPTION:
The study will a be a biologically enriched, prospectively stratified phase II trial in RAS wild type metastatic colorectal cancer patients progressing after first-line treatment with oxaliplatin, fluoropyrimidines and an anti-EGFR monoclonal antibody. Eligible patients will be prospectively allocated to either of two groups according to VEGFR2 levels (ELISA-based technique, pg/ml) at study entry.

Others angiogenetic factors levels concentration before and during treatment. VEGF, PlGF, HGF, VEGFR1, IL8, IL1a, T-cad, VEGFR3, SAP, VDBP, neuropilin1, CRP, endoglin plasma concentrations will be evaluated before each cycle according to an ELISA-based technique All patients will undergo a blood test for retrieving circulating tumor DNA (Liquid Biopsy) at selected time-points before and during treatment for determining whether the status of selected tumor biomarkers evolve during tumor progression by comparing different ctDNA samples.

All patients will receive aflibercept in combination with FOLFIRI according to the Italian label.

ELIGIBILITY:
Inclusion Criteria:

* • Histological confirmation of colorectal cancer

  * Confirmed RAS wild type patient treated with an oxaliplatin-anti EGFR treatment in 1st line
  * At least one lesion measurable with CT or MRI scan
  * Radiologically documented progression while on or after discontinuation of treatment with FOLFOX in combination with an anti-EGFR monoclonal antibody (either cetuximab or panitumumab)
  * Radiologically documented progressing disease after FOLFOX in combination with an anti-EGFR monoclonal antibody (either cetuximab or panitumumab)
  * Life expectancy plus 3 months
  * Netrophils count ³ 1.5 x 109/L
  * Platelets count ³ 100 x 109/L
  * Hemoglobin ³ 9 g/dL
  * Creatinine £ 1.5 mg/dL, Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour.Bilirubin £ 1.5 x ULN
  * AST and ALT £ 2.5 x ULN (< 5 ULN in case of liver metastases)
  * Informed written consent
  * ECOG Performance Status < 2
  * Age plus18 yrs
  * Regular follow-up feasible.
  * For female patients of childbearing potential, negative serum pregnancy test within 1 week (7 days) prior of starting study treatment,
  * Female patients must commit to using reliable and appropriate methods of contraception until at least six months after the end of study treatment

Exclusion Criteria:

* • Concomitant protocol unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),

  * Treatment with any other investigational medicinal product within 28 days prior to First Study treatment.
  * Other serious and uncontrolled non-malignant disease,
  * History or evidence upon physical examination of CNS metastasis unless adequately treated
  * Gilbert's syndrome
  * Intolerance to atropine sulfate or loperamide
  * Known dihydropyrimidine dehydrogenase deficiency
  * Treatment with CYP3A4 inducers unless discontinued > 7 days prior to First Study treatment.
  * Any of the following in 3 months prior to inclusion: grade 3-4 gastrointestinal bleeding (unless due to resected tumor), treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, or diverticulitis.
  * Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
  * Major surgery or traumatic injury within the last 28 days or until the surgical wound is fully healed whichever came later
  * Pregnant or breastfeeding women,
  * Patients with known allergy to any excipient to study drugs,
  * Bowel obstruction.
  * Uncontrolled infections
  * Known drugs or alcohol abuse
  * History of severe cardiovascular disease within 6 months prior to First Study treatment Uncontrollable hypertension, when treated with three or more drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) according to VEGFR2 levels, evaluating the difference in terms of median OS among patients with high VEGFR2 activity and patients with low VEGFR2 activity | From date of randomization until the date of death from any cause, whichever came first, assessed up to 3 years
  Overall survival time is defined as the time from inclusion to the date of death. If subject has not died, survival will be censored on the last date the subject was known to be alive (last date of follow-up)

SECONDARY OUTCOMES:
Progression free survival (PFS) defined as the interval between the start of Aflibercept-FOLFIRI therapy to tumor progression or death or last follow up visit if not progressed | time from the start of treatment untill the date of first documented progression or death from any cause, whichever came first, assessed up to 3 years
  PFS time will defined as the time of inclusion until the date of first observed disease progression or death due to any cause, if death occurs before progression is documented
Response rate (RR) defined according to the Response Evaluation Criteria in Solid Tumours (RECIST), v. 1.1 | Response of treatment is evaluated according to the RECIST criteria at the end of chemotherapyassessed up to 24 weeks
  All patients must be considered in response analysis, including those who discontinue treatment or who die for any reason prior to respnse evaluation
Toxicity Profile defined according to the Common Terminology Criteria for Adverse Events (CTCAE) v. 4.03 | every 4 cycles of chemotherapy (each cycle is 15 days), up to 16 weeks
  Treatment-emergent adverse events, drug-related adverse events and safety laboratory parameters will be analysed by CTCAE grade
Angiogenetic factors levels concentration before and during treatment. | evaluated before treatment and before each cycle (each cycle is 15 days) according to an ELISA-based technique, through completion, an overage of 1 year
  Angiogenetic factors levels concentration (VEGF, PlGF, HGF, VEGF-R, IL8, IL1a, T-cad, VEGFR3, SAP, VDBP, neuropilin1, CRP, endoglin plasma concentrations)

CONTACTS AND LOCATIONS:
Locations (16):
- Italy (16):
  - A.O. Treviglio-Caravaggio, P.le Ospedale n1, Treviglio, Bergamo
  - A.O. Humanitas Gavazzeni, Bergamo, BG
  - Policlinico Universitario D.Casula, Monserrato, Cagliari
  - A.O. Polo Oncologico Vito Fazzi, Lecce, LE
  - ASST-Rhodense, Rho, Milano
  - Istituto Clinico Humanitas, Rozzano, MI
  - AUSL di Piacenza, Piacenza, PC
  - Centro Riferimento, Aviano, PN
  - Azienda Ospedaliera San Carlo, Potenza, PZ
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Fondazione Poliambulanza, Via Bissolati 57, Brescia
  - IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Istituto Europeo di Oncologia, Milan
  - A.O.U. Policlinico di Modena, Modena
  - A.O. S.Giovanni Calabita Fatebenefratelli, Roma
  - Ospedale San Bortolo, Vicenza